CLINICAL TRIAL: NCT04581616
Title: The Effect of Ultrasound-guided Erector Spinae Block and Intraoperative Intercostal Nerve Block on Postoperative Analgesia in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202008040RINC
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia; Postoperative Pain; Ultrasound Therapy; Complications
Keywords: Erector Spinae Plane Block, ESPB; Intercostal Nerve Block, ICNB; Thoracic surgery; Postoperative pain; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICNB group (Active Comparator): After patient was turned to lateral decubitus position, local anesthetics is injected around incision site and ICNB is performed once after surgeon geys into chest cavity.
  Interventions: Procedure: Intrathoracic Intercostal Nerve Block
- ESPB group (Experimental): After patient was turned to lateral decubitus position, ESPB is performed via ultrasound guided technique before sound incision.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Intrathoracic Intercostal Nerve Block — Injection of local anesthetic into the subcostal groove, to achieve analgesia for chest region.
  Other Names: ICNB
  Arms: ICNB group
Procedure: Erector Spinae Plane Block — Injection of local anesthetic in the plane deep to the erector spinae muscles and superficial to the transverse processes, to achieve analgesia for chest region.
  Other Names: ESPB
  Arms: ESPB group

SUMMARY:
This study aims to compare the effect of ultrasound-guided erector spinae plane block and interthoracic intercostal nerve block in thoracic surgery. Interthoracic intercostal nerve block is a routine procedure during the surgery by the surgeon in our hospital, and ultrasound-guide erector spinae plane block is a relative new developed regional analgesia technique introduced since 2016 and mainly done by anesthesiologists. Both technique provide analgesic effect to some extent and reduce opiate consumption and side effects. However, no previous literature or research compare the effect of these two technique in thoracic surgery. The primary endpoint of our study is compare morphine consumption and pain score between patients undergo ESP block and patients undergo ICNB after thoracic surgery; the second endpoint is to compare the recovery condition evaluated by QoR-15 questionaire 24 hours after surgery.

DETAILED DESCRIPTION:
Sample size estimation is based on our APS team data, in which the average cumulative morphine consumption in patients underwent VATS surgery with ICNB was calculated. The mean cumulative morphine consumption was 15±8 mg of patients underwent VATS with ICNB. We assume the difference between ICNB and ESPB group reach 5 mg and aim for a power of 95 % and a risk of 0.05 for a type-1 error, at least 42 for each group needing to be recruited. 50 patients for each group, total 100 patients will be collected to avoid dropouts. Patient will be allocated to one of the trial groups using a computer-generated random number table once the consent was approved. First group is ICNB group and the second group is ESPB group.

The general anesthesia agents, induction process and routine care are the same for both groups. Once aforementioned routine cares are done, the patient will be turn into lateral decubitus position. Echo-guided ESP block will be performed after patients are turned into lateral decubitus position in ESP group; on the other side, local anesthetics will be injected at incision site and intrathoracic intercostal nerve block will be performed in ICNB group right after the surgeon makes the incision site and get into chest cavity.

Pain score (VAS) and cumulative morphine consumption will be recorded in PACU, postoperative 24H, 48H, and before discharge. Recovery condition will be evaluated via QoR-15 questionnaire in postoperative 24H, furthermore, we will follow up the patient's pain and recovery status 3 months after the operation. After collecting above data, the effect of ESP group and ICNB group on acute pain relieve, chronic pain control and recovery enhancement will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient receive thoracic surgery
* BMI between 18.5~30.0 kg.m-2

Exclusion Criteria:

* Pregnant woman
* Patient with any one of following chronic organ dysfunction: Heart failure (NYHA score =III、IV); Renal failure (eGFR< 60 ml.min-1.1.73m-2)
* Arrhythmia
* Ongoing infection or septic patient
* Chronic use of analgesic with addiction
* Coagulopathy that is not suitable for regional anesthesia performance
* Thoracic surgery that is not suitable for placement of endotracheal blocker tube
* Redo surgery

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Postoperative 48 hours
  Pain intensities in two category, namely static and dynamic, gauged by a 0-100 mm visual analogue scale, (no pain to severe pain)
Postoperative analgesic consumption | Postoperative 48 hours
  Cumulative morphine consumption in postoperative two days

SECONDARY OUTCOMES:
Recovery quality: questionnaire | Postoperative 24 hours
  Postoperative recovery quality assessed by Quality of recovery-15 (QoR-15) questionnaire, with a score range of 0-150, (poor recovery to excellent recovery)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan